CLINICAL TRIAL: NCT03178981
Title: A Pharmacokinetic Study to Examine Nicotine Delivery From E-cigarettes and a Conventional Cigarette in Healthy Subjects During a Brief Period of ad Libitum Use
Brief Title: E-cigarette Nicotine Pharmacokinetic Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: British American Tobacco (Investments) Limited (Industry)
Collaborators: LA Clinical Trials (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: BAT4217010
Record Dates: First submitted 2017-06-06; First posted 2017-06-07 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-12

CONDITIONS: Healthy Volunteers; Smoking
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Conventional cigarette (Active Comparator): Commercially-available combustible cigarette
  Interventions: Other: Use electronic cigarette or smoke conventional cigarette
- Second-generation e-cigarette A (Experimental): Prototype second-generation (closed-tank) e-cigarette
  Interventions: Other: Use electronic cigarette or smoke conventional cigarette
- Second-generation e-cigarette B (Experimental): Prototype second-generation (closed-tank) e-cigarette
  Interventions: Other: Use electronic cigarette or smoke conventional cigarette
- Second-generation e-cigarette C (Experimental): Prototype second-generation (closed-tank) e-cigarette
  Interventions: Other: Use electronic cigarette or smoke conventional cigarette
- Second-generation e-cigarette D (Experimental): Prototype second-generation (closed-tank) e-cigarette
  Interventions: Other: Use electronic cigarette or smoke conventional cigarette
- Second-generation e-cigarette E (Active Comparator): Commercially-available second-generation (closed-tank) e-cigarette
  Interventions: Other: Use electronic cigarette or smoke conventional cigarette

INTERVENTIONS:
Other: Use electronic cigarette or smoke conventional cigarette — Use of electronic cigarette or smoking conventional cigarette ad libitum for 5 minute period

SUMMARY:
This study will compare nicotine delivery and product satisfaction in healthy subjects either using several different types of electronic cigarettes or smoking a conventional cigarette.

ELIGIBILITY:
Inclusion Criteria:

1. Prior to study start, subjects must be current smokers of conventional factory-made cigarettes (eCO >10ppm at screening) who have either tried or are occasional users of e-cigarettes. Subjects must be smoking ≥10 cigarettes per day and must have done so for at least one year. Smoking status will be confirmed with a urinary cotinine level of ≥200ng/ml (determined using NicAlert cotinine test kit) and an exhaled breath CO level of >10ppm (determined using a Smokerlyzer breath CO monitor) at screening, as well as by tobacco use questionnaire.
2. Subjects will be males or non-pregnant, non-lactating females, and between 22 and 55 years of age inclusive. Age verification will be performed by checking of Federal or state-issued ID (eg. passport or driving licence) during screening.
3. Women of child-bearing potential should be using one of the following acceptable methods of contraception : combined (oestrogen and progestogen containing) oral, intravaginal or transdermal hormonal contraception associated with inhibition of ovulation; progestogen-only hormonal contraception, either oral, injected or implanted, associated with inhibition of ovulation; progestogen-only oral hormonal contraception where inhibition of ovulation is not the primary mode of action; intrauterine device (IUD); intrauterine hormone-releasing system (IUS); bilateral tubal occlusion; male or female condom with or without spermicide; cap, diaphragm or sponge with spermicide.
4. Women of non-childbearing potential may be included if they are either surgically sterile (hysterectomy and/or oophorectomy) or postmenopausal for more than 1 year and must have a negative urine pregnancy test result during screening. Women who are surgically sterile must provide documentation of the procedure by an operative report.
5. Male subjects must use an approved method of birth control during the entire study. These subjects must not donate sperm during this time.
6. Subjects must be in good health, as judged by the PI or the appropriately qualified designee based on medical history, ECG, vital signs, blood biochemistry, haematology, urinalysis and physical examination.
7. Subjects must have a body mass index (BMI) between 18 and 30 kg/m2 inclusive. Male subjects must have a weight between 60 and 120kg and female subjects between 50 and 100kg.
8. No clinically significant abnormalities in blood pressure values.
9. Subjects will have negative results for the urinary drug of abuse screening and alcohol test.
10. Subjects will have given their written informed consent to participate in the study and to abide by the study restrictions.

To be confirmed during each clinic visit:

1. Abstinence from tobacco and nicotine products will be confirmed by an exhaled breath CO reading <15ppm.

Exclusion Criteria:

1. Subjects who have a history of, or clinically active significant, neurological, gastrointestinal, renal, hepatic, cardiovascular, psychiatric, respiratory, metabolic, endocrine, haematological disease or other major disorders.
2. Subjects who have any clinically significant abnormal laboratory safety findings at Screening and prior to first product use, as determined by the PI or the appropriately qualified designee (1 repeat assessment is acceptable).
3. Subjects who have previously been diagnosed with any form of malignancy.
4. Subjects with significant allergies who in the opinion of the Principal Investigator or appropriately qualified designee should not be included.
5. Subjects who have had an acute illness (e.g. upper respiratory tract infection, viral infection, etc.) requiring treatment within 4 weeks prior to Admission.
6. Subjects who have used prescription or over-the-counter (OTC) bronchodilator medication (e.g. inhaled or oral β-adrenergic agonists) to treat a chronic condition within the 12 months prior to Admission.
7. Subjects with a recent history of or current drug or alcohol abuse who in the opinion of the Investigator should not be included. Excessive intake of alcohol within the last 6 months, defined as a regular maximum weekly intake of greater than 7 drinks for women or 14 drinks for men. One drink is defined as one pint of regular beer (5% alcohol), 200 ml of wine (12% alcohol), or 25 ml of distilled spirits (40% alcohol).
8. Subjects with an inability to communicate well with the Investigator/study staff (i.e., language problem, poor mental development or impaired cerebral function).
9. Subjects who are participating in another clinical research study or who have participated in a clinical research study in the last 2 months.
10. Subjects who have had treatment with prescription medications within 21 days or over-the-counter medication within 24 hours of the planned first product use occasion, except for those stated in the Inclusion Criteria. For all subjects, prescribed use of blood pressure (beta blockers) and lipid lowering (statin) medications are permitted.
11. Subjects who have used any drugs or substances (except tobacco) known to be strong inducers or inhibitors of any CYP enzymes (formerly known as cytochrome P450 enzymes) within a 28 days period prior to first product administration. For a list of such drugs and substances, please refer to http://medicine.iupui.edu/clinpharm/ddis/main-table/.
12. Subjects who have had any treatment with smoking cessation medications (e.g. Bupropion, Chantix or any NRT) within 30 days of the planned first product use occasion.
13. Subjects with any other clinically significant medical history, in the Investigator's opinion, including conditions which might affect drug absorption, metabolism or excretion.
14. Female subjects, who are pregnant or become pregnant during the course of the study.
15. Subjects who have lost or donated more than 450ml of blood within the 2 months preceding the first product administration.
16. Subjects who are self-reported non-inhalers (smokers who draw smoke from the cigarette into the mouth and throat but who do not inhale). Subjects who are observed as non-inhalers at Admission by the clinic staff will be excluded.
17. Subjects who are currently trying to stop smoking or to stop using e-cigarettes, or considering stopping in the next two months. All subjects will be informed that they are free to quit smoking/using e-cigarettes and withdraw from the study at any time.
18. Subjects who are unwilling or unable to comply with the study requirements.
19. Subjects who in the opinion of the Principal Investigator or their appropriately qualified designee should not participate in the study for any other reason.

To be re-confirmed during each clinic visit:

1. Subject continues to meet all screening exclusion criteria. Pregnancy test to be performed on all female subjects at each visit.
2. Receipt of any medication since screening visit that may have an impact on the safety and objectives of the study (at the Principal Investigator's discretion).

Ages: 22 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2017-06-26 (Actual); Primary Completion 2017-09-08 (Actual); Study Completion 2017-09-08 (Actual)

PRIMARY OUTCOMES:
Plasma nicotine concentration (Cmax) | -5, 1, 3, 5, 6, 7, 9, 15, 45, and 60 minutes relative to the first puff on the cigarette/e-cigarette
  Nicotine pharmacokinetics
Plasma nicotine concentration (Tmax) | -5, 1, 3, 5, 6, 7, 9, 15, 45, and 60 minutes relative to the first puff on the cigarette/e-cigarette
  Nicotine pharmacokinetics
Plasma nicotine concentration (AUC0-60) | -5, 1, 3, 5, 6, 7, 9, 15, 45, and 60 minutes relative to the first puff on the cigarette/e-cigarette
  Nicotine pharmacokinetics

SECONDARY OUTCOMES:
Number of puffs taken | During 5 minute ad libitum puffing period
Subjective measurement of product satisfaction | After 60 minute blood sampling period
Mass loss from e-cigarette cartridge during puffing | During 5 minute ad libitum puffing period

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Nides, PhD, Principal Investigator — Los Angeles Clinical Trials
Locations (1):
- Los Angeles Clinical Trials, Burbank, California, United States

IPD SHARING:
Plan to Share IPD: No